CLINICAL TRIAL: NCT04489355
Title: Assessment of Risks and Outcomes of Surgical Intervention in Patients With Ischemic Cardiomyopathy in the Early and Long-term Postoperative Period, Selection of Optimal Surgical and Surgical Treatment
Brief Title: The Effectiveness of Surgical Treatment of Patients With Ischemic Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: Tomsk NRMC ICM
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Cardiovascular Diseases; Chronic Heart Failure; Ischemic Cardiomyopathy
Keywords: Chronic heart failure; Ischemic cardiomyopathy
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Myocardial biopsy: it is planned to intraoperatively collect myocardial biopsy samples from patients with ischemic cardiomyopathy. In case of aneurysmectomy and myocardial biopsy in the middle parts of the left ventricle of the anterior, posterior, lateral walls and interventricular septum on the side of the endocardium, the wall of the aneurysm and the portion of the right atrial appendage, in the absence of an aneurysm, only the portion of the right atrial appendage.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CABG: The patients with ischemic cardiomyopathy underwent coronary artery bypass graft (CABG)
  Interventions: Procedure: coronary artery bypass graft (CABG) with surgical ventricular restoration (SVR) and mitral repair (MR)
- CABG with SVR: The patients with ischemic cardiomyopathy underwent coronary artery bypass graft (CABG) with surgical ventricular restoration (SVR)
  Interventions: Procedure: coronary artery bypass graft (CABG) with surgical ventricular restoration (SVR) and mitral repair (MR)
- CABG with mitral repair: The patients with ischemic cardiomyopathy underwent coronary artery bypass graft (CABG) with and mitral repair (MR)
  Interventions: Procedure: coronary artery bypass graft (CABG) with surgical ventricular restoration (SVR) and mitral repair (MR)
- CABG with SVR and mitral repair: The patients with ischemic cardiomyopathy underwent coronary artery bypass graft (CABG) with surgical ventricular restoration (SVR) and mitral repair (MR)
  Interventions: Procedure: coronary artery bypass graft (CABG) with surgical ventricular restoration (SVR) and mitral repair (MR)

INTERVENTIONS:
Procedure: coronary artery bypass graft (CABG) with surgical ventricular restoration (SVR) and mitral repair (MR)

SUMMARY:
The study focuses on the development of a new personalized approach to diagnostics and surgical treatment of patients with ischemic cardiomyopathy. The algorithm for selection of patients for certain type of cardiac surgery will be developed. The models for prediction of the risks and outcomes of cardiac surgery will be elaborated to reduce the rate of complications in the early and long-term postoperative period in patients with ischemic cardiomyopathy. Imaging modalities, methods for assessement of structural and functional state of the myocardium, biochemistry testing, immunohistochemical examination, and myocardial biopsy studies will be used to achieve these goals.

DETAILED DESCRIPTION:
The aim of the study is to develop a new personalized approach to diagnostics and surgical treatment of patients with ischemic cardiomyopathy.

Research Objectives:

1. To assess the prognostic values of scintigraphic indicators of myocardial perfusion, contractility, and metabolism in patients with ischemic cardiomyopathy in regard to the development of cardiac remodeling and adverse cardiovascular events in the mid term after surgery.
2. To assess the prognostic values of parameters of cardiac magnetic resonance imaging (cMRI) allowing to predict the risks of surgical intervention and chronic heart failure progression in patients with ischemic cardiomyopathy.
3. To analyze the relationships between the structural and functional state of the myocardium and the effectiveness of various types of surgery in patients with ischemic cardiomyopathy. The structural and functional state of the myocardium is assessed by the instrumental methods including myocardial scintigraphy, cMRI, stress echocardiography, spiroergometry, and intraoperative fluometry.
4. To identify the myocardial biopsy-based predictors of adverse outcome in patients with ischemic cardiomyopathy in the early and mid term postoperative period in patients with ischemic cardiomyopathy.
5. To study the relationships between tissue and molecular biomarkers, severity of ischemic cardiomyopathy, and the outcomes in patients with ischemic cardiomyopathy in the postoperative period.
6. To introduce new and to optimize existing methods of surgical treatment in patients with ischemic cardiomyopathy.
7. To develop an algorithmic model for assessing the risks and predicting outcomes of surgical intervention in patients with ischemic cardiomyopathy in the postoperative period.

Methods:

1. Clinical status of the patient: collection of complaints, medical history, physical examination, assessment of anthropometric indicators (measurement of body weight, height, BMI), and demographic indicators before and in the control period after surgical treatment.
2. General clinical examination: standard 12-lead ECG, general urine analysis, general blood analysis, blood chemistry, coagulation, chest x-ray, ultrasound of the carotid and femoral arteries.
3. Echocardiography: determination of the type of aneurysm according to Di Donato; measuring the distance between the papillary muscles of the left ventricle; assessing the depth of co-optation of the mitral valve cusps; measuring Vena contracta; measuring the radius of the proximal regurgitation zone, cm; Effective Regurgitant Orifice Area (EROA, cm2); assessing systolic index and sphericity index. Stress echocardiography with dobutamine. Before stress echocardiography on a Vivid E9 ultrasound system (GE, Healthcare), continuous intravenous administration of dobutamine HEXAL, starting from 5 μg/kg/min and increasing its dose every 3 minutes to 10, 15, 20, 30, and 40 μg/kg.
4. Coronarography for assessing the anatomy and condition of the coronary pool using an angiographic unit (Axiom Artis/Innova 2121-IQ (General Electric, USA)).
5. Contrast-enhanced cMRI to assess the following parameters:

   * mass of viable left ventricular myocardium;
   * volumes of cardiac cavities;
   * diameter of the mitral and tricuspid valve rings with the determination of regurgitation degree;
   * the long axis of the ventricle;
   * left ventricular ejection fraction;
   * visualization of akinetic and hypokinetic myocardium;
   * the presence of blood clots in the cavities of the heart;
6. Six-minute walk test.
7. Spiroergometry by SCHILLER complex with a GanshornPowerCube gas analyzer.
8. Determination of the plasma and serum levels of the NT-proBNP, endothelin-1, troponin I, galectin-3, ST-2, matrix metalloproteinases (MMP) 2 and 9, and C-reactive protein.
9. Evaluation of myocardial perfusion by single-photon emission computed tomography using radiopharmaceuticals 199 Tl chloride or 99m Tc. Myocardial perfusion scintigraphy with Tc-methoxyisobutylisonitrile (99mTc-MIBI) and iodine-123-labeled iodine-123-phenylmethylmethylene diode and metabolic scintigraphy with 123I-FMPDKc. Stress ventriculography with 99-Tc-pyrophosphate by GKS-301T gamma camera (VNIIMP-VITA, Russia).
10. Intraoperative fluometry of coronary grafts during coronary artery bypass grafting using the Medistim VeriQ System.
11. Myocardial biopsy: it is planned to take myocardial biopsy samples in patients with ischemic cardiomyopathy intraoperatively. In case of aneurysmectomy, myocardial biopsy will be sampled in the middle left ventricular (LV) parts of the anterior, posterior, lateral walls and the endocardium, the wall of the aneurysm and the portion of the right atrial appendage, the right atrial appendage in the absence of aneurysmectomy. The preparation of histological samples will be carried out in a standard way: fixation of biopts in formalin with further filling in a paraffin medium and staining with hematoxylin and eosin with determination of morphometric indicators. For histochemical reactions, biopsy samples freshly frozen in liquid nitrogen will be used. The enzymatic activity of succinant dehydrogenase (LDH), lactate dehydrogenase (LDH), and 3-hydroxybutyrate dehydrogenase (3-HBDH) will be studied using the Lojda tetrazolium method according to the intensity of staining of the structure using the ImageJ program (NIH, USA).
12. Statistical processing of data:

Structured collection of patient data will be performed in a database formed on the platform of the Microsoft Excel 2010 software (Microsoft Corp., USA). Statistical processing of the results will be carried out using the SPSS 23.0 for Windows software package (IBM Corp., Armonk, NY, USA). The normality of the law of distribution of quantitative indicators will be checked using the Shapiro-Wilks criterion. Normally distributed parameters will be presented as mean value (M) and standard deviation (StD) in the form M ± StD; not normally distributed parameters will be presented as median (Me) and the 1st and 3rd interquantile intervals (Q25 - Q75) in the form of Me [Q25; Q75]. Qualitative data will be described by the frequency of occurrence or its percentage. To find statistical dependences, to determine their strength and direction, the Pearson correlation coefficient (r) (for normally distributed parameters) and Spearman correlation coefficient (for for not normally distributed parameters and for qualitative indicators in the ordinal scale) will be calculated. Using logistic regression, significant predictors will be identified for the values of reverse remodeling in the long term after surgical treatment. When conducting a multivariate analysis of interconnections, first, by means of a univariate analysis, the main parameters that influence the studied value will be identified, then, based on the search for intergroup correlations, the signs that have a moderate or strong relationship will be eliminated, and multivariate modeling of the relationships will be performed.

Survival analysis will be performed using the Kaplan-Meier method. All statistics will be considered significant at p <0.05.

During the work, the methods of statistical analysis can be revised and (or) supplemented.

ELIGIBILITY:
Inclusion Criteria:

* left ventricular ejection fraction less than or equal to 40%; a history of myocardial infarction with a duration of more than 3 months and/or stenosis of more than 75% of the trunk of the left coronary artery, or proximal stenosis of the anterior descending artery and/or stenosis of more than 75% of two or more coronary arteries; final LV systolic index greater than or equal to 60 ml / m2 according to echocardiography, age 18-70 years

Exclusion Criteria:

* the presence of organic heart defects of rheumatic and infectious etiology; acute myocardial infarction; less than 3 months after acute coronary or cerebrovascular events; severe pulmonary hypertension not associated with mitral regurgitation (above 75 mmHg); contraindications for operations with cardiopulmonary bypass; chronic alcoholism (including alcoholic damage to the heart), mental disorders; severe course of bronchial asthma, chronic obstructive pulmonary disease in the acute stage; oncological diseases in the terminal stage, refusal of the patient or relatives to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic cardiomyopathy with indications for cardiac surgery
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2013-01-28 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with postoperative left ventricular remodeling according to echocardiography. | 12 months
  Number of participants with a decrease in left ventricular end-systolic volume by 15% or more.
Cardiac death | 12 months
  Cardiac death, %

SECONDARY OUTCOMES:
Number of participants with increased exercise tolerance | 12 months
  Number of participants with increased exercise tolerance according to spiroergometry by 15% or more.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir M Shipulin, MD, PhD, Study Chair — Cardiology Research Institute, Tomsk NRMC
Locations (1):
- Tomsk National Research Medical Center of the Russian Academy of Sciences, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (text, tables, figures, and appendices), underlying the results of the trial, will be shared with researchers to achieve the aims in the approved proposal.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Proposals may be submitted up to 36 months following publication of the results of the trial. After 36 months, the data will be available in the Center's data ware house but without investigator support other than deposited metadata.
Access Criteria: Information regarding submitting proposals and accessing data may be requested from the principal investigator by e-mail.